CLINICAL TRIAL: NCT00348088
Title: CXCL1 Biomarker Study in Metastatic Melanoma
Brief Title: Melanoma Biomarker Study
Status: Completed | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: J05122; NA_00001940
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Metastatic Melanoma
Keywords: Metastatic; Melanoma; Untreated; Biomarker
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to measure the level of a specific protein, CXCL1, in the blood of patients with untreated, metastatic (Stage IV) melanoma. These levels will be compared to blood levels in normal controls. If the levels are elevated in metastatic melanoma, further studies to determine if this correlates with presence and extent of disease will be pursued.

DETAILED DESCRIPTION:
Malignant Melanoma has rapidly increased in incidence over the past thirty years, at a rate of roughly 3% per year. In 2005, approximately 59,000 new cases of melanoma were diagnosed with 8000 deaths. While the majority of early melanomas can be surgically cured, advanced melanoma has an extremely poor prognosis. Current chemotherapy and immunotherapy options for advanced melanoma still offer response rates of only 10-20%. Thus, the elucidation of biomarkers in melanoma, both diagnostic and prognostic, is an important area for investigation.

CXCL1 is a chemokine whose expression is upregulated in melanoma. We postulate that CXCL1 plays an important role in the progression of melanoma to invasive disease. Our hypothesis states that serum CXCL1 levels correlate with the presence of melanoma.

Aims:

1. To measure serum levels of CXCL1 in untreated, metastatic melanoma patients and to compare to serum CXCL1 levels in normal controls.
2. To measure and compare centrally and peripherally collected serum CXCL1 levels in untreated, metastatic melanoma.

Blood will be collected from metastatic melanoma patients on one occasion, both peripherally and centrally. Control will have blood collected peripherally on one occasion. The blood will be processed and then tested in a blinded, batched fashion.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic diagnosis of melanoma; primary may be cutaneous, mucosal or ocular.
2. Evidence of metastatic disease based on standard AJCC staging.
3. Willing to give written informed consent.
4. Willing and able to comply with protocol procedures.
5. At least 18 years of age.
6. No prior chemotherapy, immunotherapy, or radiotherapy.
7. Are able to safely donate 50 mL of blood.
8. Have a central venous catheter in place (this will not be placed for participation in this trial)

Exclusion Criteria:

1. Known diagnosis of a chronic inflammatory disease, ie: Rheumatoid Arthritis, Systemic Sclerosis, Inflammatory bowel disease
2. Known diagnosis of NYHA class 3 or 4 Congestive Heart Failure
3. Are unable to safely donate 50 mL blood
4. Known HIV, Hepatitis B, or Hepatitis C infection.
5. Any malignancy within 5 years, other than melanoma (for patients); Have any malignancy within the past 5 years including melanoma (for normal controls). Basal cell and squamous cell skin cancers are permitted in all participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Malignant Melanoma
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2006-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Observational study only | May 2006-September 2011
  To determine, via sandwiched ELISA, the presence and level of CXCL1 in the serum of patients with metastatic melanoma and to compare these values with CXCL1 levels in normal controls.

SECONDARY OUTCOMES:
Observational study only | May 2006-September 2011
  To compare serum CXCL1 levels collected peripherally and centrally, in metastatic melanoma patients and To collect serum samples for future study.

CONTACTS AND LOCATIONS:
Overall Officials: William H Sharfman, MD, Principal Investigator — Johns Hopkins University Sidney Kimmel Comprehensive Cancer Center
Locations (1):
- Johns Hopkins University - Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States